CLINICAL TRIAL: NCT06050447
Title: Factors Affecting the Results of Treatment of Patients With Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Immanuel Kant Baltic Federal University (Other)
Collaborators: Center of Endourology "Endocenter" (Other)
Responsible Party: Sponsor
Other Study IDs: 5995465480
Record Dates: First submitted 2023-08-28; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectal Cancer; Colorectal Adenocarcinoma; Colorectal Neoplasms Malignant; Rectal Adenocarcinoma
Keywords: Colorectal cancer; Rectal cancer; Colon cancer; Colorectal surgery; anastomotic leakage; postoperative complications; recurrence rate; cancer-specific survival; recurrence-free survival
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Anastomotic Leak; Postoperative Complications | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with right-sided colon cancer: Tumors located anywhere from the cecum to the proximal transverse colon.
  Interventions: Procedure: Right hemicolectomy
- Patients with left-sided colon cancer: Tumors located anywhere from the distal transverse colon to the rectosigmoid junction
  Interventions: Procedure: Left hemicolectomy; Procedure: Sigmoid colon resection
- Patients with rectal cancer: Tumors located in rectosigmoid junction and in the rectum with/without the external sphincter or the levator muscles invasion
  Interventions: Procedure: Anterior resection of the rectum; Procedure: Low anterior resection of the rectum; Procedure: Abdominoperineal resection
- Patients with right- and left-sided colon cancer (primary multiple cancer): Patients with primary multiple cancer tumors
  Interventions: Procedure: Total Colectomy

INTERVENTIONS:
Procedure: Right hemicolectomy — Resection of the caecum and ascending colon is appropriate for patients with tumors located anywhere from caecum to the transverse colon
  Groups: Patients with right-sided colon cancer
Procedure: Left hemicolectomy — Resection of the sigmoid colon is appropriate for patients with tumors located anywhere from the distal transverse colon to the rectosigmoid junction.
  Groups: Patients with left-sided colon cancer
Procedure: Sigmoid colon resection — Resection of the sigmoid colon is appropriate for patients with tumors located in the sigmoid colon
  Groups: Patients with left-sided colon cancer
Procedure: Anterior resection of the rectum — AR is appropriate for tumors located in rectosigmoid junction and in the proximal rectum
  Groups: Patients with rectal cancer
Procedure: Low anterior resection of the rectum — LAR is appropriate for tumors located in the middle and low rectum
  Groups: Patients with rectal cancer
Procedure: Abdominoperineal resection — APR is appropriate for distal rectal cancers that invade the external sphincter or the levator muscles
  Groups: Patients with rectal cancer
Procedure: Total Colectomy — Total abdominal colectomy may be indicated for patients with primary multiple cancer tumors
  Groups: Patients with right- and left-sided colon cancer (primary multiple cancer)

SUMMARY:
The study attempts to quantify the relative risks for mortality, anastomotic leakage and other early and late postoperative complications, recurrence rate, cancer-specific survival, recurrence-free survival after colorectal surgery for patients with colorectal cancer depending on the localization of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary adenocarcinoma of bowel;
* All patients who have indications for surgical treatment of colorectal cancer based on the decision of the oncological council;
* Signed informed consent with agreement to attend all study visits;

Exclusion Criteria:

* Unresectable tumor or contradictions to surgery;
* Indications for chemotherapy or radiation therapy prior to surgery;
* Patient withdrawal from the trial or loss of follow-up;
* Emergent operation;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An unselected, consecutive regionwide cohort during 3 years, with a 3-year follow-up
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate | 3 months after surgery
  Anastomotic leakage rate after colorectal resection.
  AL is confirmed by one or more of the following conditions:
  * fecal discharge from the pelvic drainage at any time after surgery
  * rectovaginal fistula defined as fecal or mucus discharge from the vagina
  * pelvic sepsis as defined by the collection of pus/ fecal material in the pelvis documented by CT scan
  * contrast present outside of the anastomosis as seen by X-Ray contrast enema proctography or CT contrast enema proctography
Mortality rate | 3 years after surgery
  the overall mortality after colorectal cancer surgery

SECONDARY OUTCOMES:
30-day complication rate | 30 days after surgery
  The number of patients with complications after colorectal resection. All complications will be assessed according to the Clavien-Dindo classification. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V).
  Grade I - Any deviation from the normal postoperative course without the need for treatment.
  Grade II - Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III - Requiring surgical, endoscopic or radiological intervention
  * IIIa - Intervention not under general anesthesia
  * IIIb - Intervention under general anesthesia Grade IV - Life-threatening complication requiring IC/ICU-management
  * IVa - single organ dysfunction (including dialysis)
  * IVb - multiorgandysfunction Grade V - Death of a patient
Recurrence rate | 3 years after surgery
  All cases of colorectal cancer recurrence
Cancer-specific survival | 3 years after surgery
  The number of patients survived within 3 years after the diagnosis
Recurrence-free survival | 3 years after surgery
  The number of patients without cancer recurrence within 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail A Agapov, PhD, Principal Investigator — Baltic Federal University
Locations (1):
- Baltic Federal University, Kaliningrad, Kaliningrad Oblast, Russia

IPD SHARING:
Plan to Share IPD: No